CLINICAL TRIAL: NCT01619397
Title: A Clinical Investigation to Evaluate In-use Genital Tolerance and User Acceptability of a Xanthan Gum Coating on a Standard Natural Rubber Latex Condom in Healthy Volunteer Mutually Monogamous Adult Couples
Brief Title: Evaluation of Tolerance and Acceptability of a Coated Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NPD 684_03
Record Dates: First submitted 2012-06-01; First posted 2012-06-14 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Tolerance and Acceptability of a New Condom Coating
Keywords: Condom; Medical Device

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Condom (Other): Test condom with new Xanthan gum condom coating
  Interventions: Device: Test condom with new Xanthan gum condom coating

INTERVENTIONS:
Device: Test condom with new Xanthan gum condom coating

SUMMARY:
This Clinical Investigation is designed to provide tolerance, acceptability and safety data of a new condom coating, in its intended use to support future application for CE Mark.

DETAILED DESCRIPTION:
The Investigational Device is a standard Natural Rubber Latex (NRL) condom with a coating on the inside and outside. The Investigational Device is dry to the touch on removal from the foil. When the coated condom comes into contact with body fluids upon penetration it absorbs the moisture and forms a lubricious (slippery) layer on the condom. From this point, the coating and the standard NRL condom feel and behave like a standard pre lubricated condom.

Condoms are a widely used, cheap and effective contraceptive and an important primary prevention strategy that can substantially reduce the likelihood of transmitting sexually transmitted infections (STI's) (Holmes et al, 2004). Consumer studies have revealed that the 'messiness' associated with pre lubricated condoms can be off putting to the consumer and possibly deter use completely. It is thought that as the condom coating is initially dry to the touch this may remove the 'messiness'.

The duration of the Investigation is 3 days. In that time subjects will attend the clinic 3 times, (Day 1, Day 2 and Day 3) for baseline assessments and subsequent Clinical Assessments. Clinical Assessments will include an examination of the external genitals (both male and female subjects) and internal genitals (female subjects only) in order to make an assessment of dermal tolerance of the area when exposed to a Project Unusual Condom in-use.

Couples will be provided with Investigation Device at visit 1 and Visit 2. There is a 24 hour period after receipt of Investigational Device in which couples are asked to use the condom for 1 act of vaginal intercourse, recording compliance and their experience of the Investigational Device in a Diary Card and questionnaire.

Assessments of tolerance will be made by the PI throughout the Investigation. The PI is a Physician with extensive Dermatology training. Assessments of dermal tolerance will include scoring particular sites according to a Total Irritancy score, providing a Global Assessment of Tolerance and at the end of the Clinical Investigation the Investigator will make an Overall Tolerance Rating Statement.

ELIGIBILITY:
Inclusion criteria:

* Healthy sexually active mutually monogamous heterosexual couples.
* Subjects at least 18 years of age
* Subjects who are willing and able to take part, attend all required visits, able to understand the information given to them and give written consent
* Couples who are be experienced latex condom users as defined by repeated use without significant problems.
* Couples must agree to use the condoms provided plus be using one other acceptable form of non barrier contraception (i.e. sterilisation/vasectomy, intra-uterine device (IUD) or intra-uterine system (IUS), hormonal contraception) unless female partner is post-menopausal (i.e. over 50 and, prior to screening, amenorrhea for at least 12 months after cessation of exogenous hormone treatment) in which case no second form of contraception is required.
* No signs of abnormalities in the medical history that the investigator would consider as clinically relevant.
* No clinically relevant findings in physical assessments
* Subject not aware of any reason why they will not be able to engage in 1 act of vaginal intercourse per Condon Use Period.

Exclusion Criteria:

* Presence or history of allergy or sensitivity to topical vaginal products Latex, Xanthan Gum or any other Investigation products
* Pre-existing skin or systemic allergic reaction or severe eczema
* Previous history of frequent problems associated with the use of condoms
* Currently active or a history of recurrent STI's including HIV infection in one or either partner.
* Participation in a clinical trial in the previous month which could, in the opinion of the investigator, affect the outcome of the Investigation.
* Intentions to continue use of concurrent vaginal lubricants or treatments for the duration of the Investigation.
* Either partner with genital piercing
* Female partners who are pregnant or breast feeding
* Female partners seeking to become pregnant in the duration of the Investigation
* Female partner who has been diagnosed with or treated for a vaginal complaint in the previous 3 months which in the Investigators opinion indicated the partner is unsuitable for the Investigation
* Female partner suffering from known vaginal dryness
* Female partner using medication which would affect vaginal mucosal secretion, such as Chlorpheniramine.
* Male partners using medication that would affect ability to obtain and maintain an erection through to normal ejaculation
* Male partners with abnormal penile anatomy that would affect ability to keep condom in place during intercourse
* Males partner with diagnosis of penile skin condition within previous 3 months (e.g. conditions associated with balanoposthitis: penile psoriasis; lichen sclerosis; eczema) as confirmed by subject and by genital examination.
* Intentions to continue to use antihistamines, anti inflammatory drugs, or pain killers for the duration of the Investigation
* Suffering from any condition which could, in the opinion of the Investigator, affect the outcome of the Investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
To demonstrate dermatological tolerance. | The active phase of this Investigation lasted less than 1 week per participating couple and within this period there were a total of 3 visits (Day 1, Day 2 and Day 3).
  To determine the in-use genital tolerance of Xanthan gum coating on a standard natural rubber latex (NRL) condom, as a lubricant for vaginal intercourse

SECONDARY OUTCOMES:
User acceptability. | The active phase of this Investigation lasted less than 1 week per participating couple and within this period there were a total of 3 visits (Day 1, Day 2 and Day 3).
  To assess user acceptability of Xanthan gum coating on standard NRL condom as defined by 70% of subjects selecting the top two boxes in applicable questions of acceptability questionnaire.
Assessment of safety profile. | The active phase of this Investigation lasted less than 1 week per participating couple and within this period there were a total of 3 visits (Day 1, Day 2 and Day 3).
  To determine in-use safety of Xanthan gum coating on standard NRL condom in terms of frequency and severity of device deficiencies, malfunction, or adverse device effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Alba Science Ltd, 24 Brought Street, Edinburgh, United Kingdom